CLINICAL TRIAL: NCT04905992
Title: Is a Single Daily Session Combining Hypertonic Saline Nebulisation and Airway Clearance Techniques Sufficient to Obtain Long-term Clinical Benefits in People With Bronchiectasis? A Randomised Non-inferiority Trial.
Brief Title: Is a Single Daily Session Combining HS + Physio Sufficient to Obtain Long-term Clinical Benefits in Bronchiectasis?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Clínico Universitario Lozano Blesa (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Universidad San Jorge (Other)
Responsible Party: Principal Investigator, Beatriz Herrero-Cortina, PhD Beatriz Herrero Cortina, Hospital Clínico Universitario Lozano Blesa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HS_nonInferiority
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Bronchiectasis; Airway Clearance Impairment
Keywords: Airway clearance techniques; Hypertonic saline; Hyperosmolar agents; Oscillating positive expiratory pressure
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Intervention Model Description: A non-inferiority randomized clinical trial (single-blinded assessor).
Who Masked: Outcomes Assessor
Masking Description: The assessors in charge of the measures will be blind to the group assignment of participants until the study has been completed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single daily session (Hypertonic saline + airway clearance techniques) (Experimental): The experimental group will perform a daily session at home including nebulisation of 5 mL of hypertonic saline (at 6%) followed by 15 min of airway clearance techniques (oscillating positive expiratory pressure therapy) for 6 months.
  Interventions: Other: Hypertonic saline at 6%; Other: Airway clearance techniques (oscillating positive expiratory pressure therapy)
- Twice daily session (Hypertonic saline + airway clearance techniques) (Active Comparator): The control group will perform two daily sessions at home involving nebulisation of 5 mL of hypertonic saline (at 6%) followed by 15 min of airway clearance techniques (oscillating positive expiratory pressure therapy) for 6 months.
  Interventions: Other: Hypertonic saline at 6%; Other: Airway clearance techniques (oscillating positive expiratory pressure therapy)

INTERVENTIONS:
Other: Hypertonic saline at 6% — Participants will start the sessions by inhaling a short-acting bronchodilator or an anticholinergic to avoid the presence of bronchospasm during nebulisation. The hypertonic solution (at 6%) will be administered through the Turbo Boy nebuliser (Pari®). The intervention will take place at home.
Other: Airway clearance techniques (oscillating positive expiratory pressure therapy) — Following nebulisation, participants will perform airway clearance techniques using an oscillating positive expiratory pressure device for at least 15 minutes. The intervention will take place at home

SUMMARY:
The present study will aim to find out whether a home treatment in people with bronchiectasis consisting of a single daily session to facilitate expectoration (combining nebulization of hypertonic saline (HS) at 6% followed by airway clearance techniques) is at least as effective as performing two sessions per day following the same process in each of the sessions, during a period of 6 months.

DETAILED DESCRIPTION:
A non-inferiority randomised clinical trial (single-blind) will be conducted. At least 50 participants will be recruited from the outpatient clinics of the Hospital Clinic in Barcelona and the Clinical University Hospital in Zaragoza. The experimental group will nebulize once/day the hypertonic saline (HS) solution followed by airway clearance exercises (15 min) for 6 months. The control group will follow the same procedure, but the frequency of the sessions will be twice a day (reference as usual clinical practice). The main study outcomes will be: (1) cough severity (primary endpoint), symptoms and quality of life; (2) functional exercise capacity; (3) time to first exacerbation and total number of exacerbations; (4) indirect measures of mucociliary transport (rheology and concentration of solids in sputum samples); (5) inflammatory parameters; (5) tolerance, safety and adherence to treatment. Measurements will be taken at baseline (prior to randomization), at 1 month, 3 months, and 6 months. Finally, hypothesis testing will be performed using a linear mixed model (2x3) of repeated measures, establishing a priori a margin of non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. a total score less than 16 on the Leicester Cough Questionnaire
3. chronic daily expectoration over at least 3 months
4. being in a period of clinical stability during the previous 4 weeks
5. presenting a forced expiratory volume in 1 second (FEV1) value greater than 40% of predicted or >1 L
6. obtaining informed consent.

In addition, all participants will have had to satisfactorily pass the tolerability tests, which will be performed twice: i) on the first day; ii) and the following week.

Exclusion Criteria:

1. having received nebulised mucoactive treatment during the previous year
2. frequent haemoptysis (≥ 2 times/month)
3. diagnosis or suspicion of cystic fibrosis by genetic study or sweat test
4. being under active treatment for nontuberculous mycobacteria (NTM)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Impact of coughing on quality of life | 6 months after starting the intervention
  The Leicester Cough Questionnaire (LCQ) will be used to assess the daily cough impact

SECONDARY OUTCOMES:
Impact of coughing on quality of life | Baseline point, 1 month and 3 months after starting the intervention
  The Leicester Cough Questionnaire (LCQ) will be used to assess the daily cough impact
Disease-specific quality of life questionnaire | Baseline point, 1 month, 3 months and 6 months after starting the intervention
  The Quality of life of Bronchiectasis (QoL-B) questionnaire will be used to evaluate the quality of life
Disease-specific symptoms questionnaire | Baseline point, 1 month, 3 months and 6 months after starting the intervention
  The Bronchiectasis Impact Measure (BIM) outcome measure will be used to analyse the symptoms
Exercise capacity | Baseline point, 1 month, 3 months and 6 months after starting the intervention
  The sit to stand test (1 minute) will be used to assess the exercise capacity
Exercise capacity | Baseline point
  The six minute walk distance (6MWT) will be used to assess the exercise capacity
Exacerbations | From baseline point to the end of the intervention (6 months)
  The number of exacerbations, the severity of exacerbations (hospital admission) and the time to the first exacerbation will be recorded prospectively
Biophysical properties of spontaneous sputum samples | Baseline point, 1 month, 3 months, 6 months
  Spontaneous sputum samples will be collected to analyse the main biophysical markers
Inflammation markers (airway inflammation and systemic inflammation) | Baseline point, 1 month, 3 months, 6 months
  Blood and salivary samples will be collected to analyse the main inflammatory markers (neutrophil elastase, cytokines, peptides)

OTHER OUTCOMES:
Lung Function | Baseline point, 1 month, 3 months, 6 months
  Forced spirometry (forced expiratory volume in 1 second [FEV1] and forced vital capacity [FVC]) will be perform for safety analysis following the American Thoracic Society / European Respiratory Society guidelines
Adverse events during sessions | Baseline point, 1 month, 3 months, 6 months
  Adverse events during nebulisation period will be recorded using a Likert scale and participants will also complete the Self-Reported Medication Scale

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Alcaraz-Serrano, Principal Investigator — Hospital Clinic of Barcelona; Beatriz Herrero-Cortina, Principal Investigator — Hospital Clínico Universitario Lozano Blesa
Locations (2):
- Spain (2):
  - Hospital Clinic, Barcelona
  - Beatriz Herrero Cortina, Zaragoza

IPD SHARING:
Plan to Share IPD: No